CLINICAL TRIAL: NCT06132139
Title: VisAR Augmented Reality Navigation of Ventriculostomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Hong, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY02002144
Record Dates: First submitted 2023-09-21; First posted 2023-11-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Hydrocephalus; Subarachnoid Hemorrhage; Brain Trauma
MeSH Terms: conditions — Hydrocephalus; Subarachnoid Hemorrhage; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VisAR Navigation (Experimental): Patients randomly assigned to this arm will have their EVD placed using VisAR navigation.
  Interventions: Device: VisAR
- Freehand Navigation (No Intervention): Patients randomly assigned to this arm will have their EVD placed using freehand navigation, the typical standard of care.

INTERVENTIONS:
Device: VisAR — The study device is a Microsoft HoloLens which uses Novarad's proprietary software and is collectively known as VisAR.
  Arms: VisAR Navigation

SUMMARY:
This study is intended to evaluate the feasibility of using VisAR augmented reality surgical navigation during placement of an external ventricular drain (EVD). The investigators are interested in confirming the design of the VisAR headset is compatible with this bedside procedure.

DETAILED DESCRIPTION:
A secondary objective of this study is to compare the accuracy of freehand EVD navigation, the current standard of care, with VisAR augmented reality surgical navigation. The intent is to demonstrate the advantages to the patient by the use/application of this next generation navigation technology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years and older, determined to need an external ventricular drain (EVD) or ventriculostomy catheter by the attending neurosurgeon secondary to a variety of pathologies, including obstructive hydrocephalus, trauma and subarachnoid hemorrhage.

Exclusion Criteria:

* Patients less than 18 years of age.
* Pregnant women.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Determining navigation system accuracy based on anatomical location and Kakarla scoring system. | During surgery
  The accuracy of VisAR in placement of EVDs primary assessment will be graded based on the anatomical location of the EVD, known as the Kakarla scoring system. The Kakarla scoring system has 3 grades of accuracy of placement based on the location of the catheter tip.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hong, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center